CLINICAL TRIAL: NCT02373657
Title: Water Uptake for Health in Amhara Pilot
Acronym: WUHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10-02169-B
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Trachoma
Keywords: trachoma; soil transmitted helminths; water; hand washing
MeSH Terms: conditions — Trachoma | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WASH Intervention (Experimental): In these seven communities we built a well in a central location for all state team residents. We plan on providing "tippy-taps" (water and soap dispensers), instruction in soap-making, and hygiene education to these communities. We will also put fly traps in the communities to see if wells reduce flies. We plan on performing monitoring visits at 12 months and 24 months, in order to assess clinically active trachoma, ocular chlamydia infection, nasopharyngeal macrolide resistance, soil transmitted helminths, and childhood growth (height and weight). We will also perform assessments of the adequacy of the intervention, by conducting household surveys to assess hygiene behavior, access to water and latrines, and fly density.
  Interventions: Behavioral: instruction in soap-making and hygiene education
- Control (No Intervention): In these seven communities, we plan to perform monitoring visits at 12 months and 24 months, in order to assess clinically active trachoma, ocular chlamydia infection, nasopharyngeal macrolide resistance, soil transmitted helminths, and childhood growth (height and weight). We will also perform assessments of the adequacy of the intervention, by conducting household surveys to assess hygiene behavior, access to water and latrines, and fly density.

INTERVENTIONS:
Behavioral: instruction in soap-making and hygiene education
  Arms: WASH Intervention

SUMMARY:
Trachoma is a blinding disease caused by ocular strains of Chlamydia trachomatis. The Carter Center and Proctor Foundation have been jointly conducting trachoma research in the Goncha Siso Enese woreda of Amhara for the past 8 years, through a series of clinical trials. We have found that repeated mass administration of oral azithromycin can greatly reduce the prevalence of trachoma, but mass antibiotics have been unable thus far to eliminate infection. The World Health Organization recommends not only antibiotics for control of trachoma, but an entire SAFE strategy (Surgery for in-turned eyelids, Antibiotics, Facial hygiene promotion, and Environmental improvements such as latrines and water points). Trachoma is more common in villages and households with poor access to water and latrines, so improving the public health infrastructure is thought to be important for limiting transmission of trachoma. However, there is very little evidence to support the efficacy of installing new water points for trachoma. There has been only one previous attempt to study the role of hand dug well installation for trachoma control, and this study, conducted in Niger, found that installing wells was not effective. We now propose a project to improve the public health infrastructure of Goncha Siso Enese woreda by helping with the construction of water points (e.g., hand-dug wells) and providing hygiene education, in order to determine whether improving access to water and hygiene information will be effective for control of trachoma and soil-transmitted helminths.

ELIGIBILITY:
Inclusion Criteria:

* All residents residing in the state-teams which are randomly selected for this study.

Exclusion Criteria:

* Refusal of village chief (for village inclusion), or refusal of parent or guardian (for individual inclusion)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4068 (Actual)
Dates: Start 2014-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of ocular chlamydia infection (0-5 year olds) | 24 months
Nasopharyngeal macrolide resistance (0-5 year olds) | 24 months
Prevalence of soil transmitted helminths (Ascaris, Trichuris trichiura, and hookworm) (0-5 year olds) | 24 months

SECONDARY OUTCOMES:
Childhood growth (weight controlled for height among children aged 0-5 years at baseline) | 24 months
Clinically active trachoma in children aged 0-5, as determined by the WHO simplified grading system | 24 months
Prevalence of enteric viruses using PCR (0-5 year olds) | 24 months
Self report childhood morbidity | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Keenan, MD, MPH, Principal Investigator — F.I. Proctor Foundation, University of California San Francisco
Locations (1):
- The Carter Center, Addis Ababa, Ethiopia